CLINICAL TRIAL: NCT04041817
Title: Pulmonary and Ventilatory Effects of Trigger Modulation in Intubated ICU Patients Spontaneously Breathing With Pressure Support Ventilation. A Physiopathology Exploratory Study.
Brief Title: Pulmonary and Ventilatory Effects of Trigger Modulation in Intubated ICU
Acronym: Trigger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trigger - RBHP 2018 GODET; 2018-A03307-48 (Other: ANSM)
Record Dates: First submitted 2019-07-25; First posted 2019-08-01 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: ICU Patients; Intubation; Spontaneously Breathing; Pulmonary Function; Tracheotomy
Keywords: ICU; Pressure support ventilation; Spontaneous breathing; Trigger; Weaning of mechanical ventilation

STUDY DESIGN:
Masking Description: Statistical analysis will be conducted by an independant statistician not involved in data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trigger increasing steps (Experimental): Trigger variations will be performed following increasing steps of 2 L/min every 15 minutes. End expiratory lung volume and lung aeration will be conducted using elecrical impedance tomography. Diaphragmatic motion and thickening will be analyzed by ultrasonography. Work of breathing will be evaluated using gastric and oesophageal pressure measurements.
  Measurements will be conducted during the last minute of each step.
  Interventions: Other: Trigger setting of pressure support ventilation

INTERVENTIONS:
Other: Trigger setting of pressure support ventilation — Trigger variations will be performed following increasing steps of 3 L/min every 15 minutes, from 0.2 to 15 L/min (0.2 - 3 - 6 - 9 - 12 - 15).

SUMMARY:
Pressure support ventilation allows intubated ICU patients to breathe spontaneously. Among specific settings, the adjustment of the trigger value (or threshold for triggering the ventilator) has not been explored to date. The trigger threshold corresponds to the sensitivity of the ventilator to detect patient's inspiratory effort and then deliver the predefined pressure support to inflate the lungs and deliver a tidal volume. The purpose of this study is to explore the influence of trigger level on pulmonary and ventilatory physio (-patho)logical parameters in spontaneously breathing ICU patients.

DETAILED DESCRIPTION:
The use of invasive mechanical ventilation is one of the most frequent therapies in intensive care units (ICUs). There are several types of indications, depending on the failure: essentially neurological, hemodynamic or respiratory.

In recent years, the notion of lung damage induced by mechanical ventilation (VILI) has led to major changes in ventilator settings in both ICUs and operative rooms (Ors). The reduction of the tidal volume (TV) to 6-8 mL/kg of ideal body weight, the use of an individualized positive end-of-expiratory pressure (PEEP) and the possible use of pulmonary aeration optimization therapies (alveolar recruitment manoeuvres, prone positioning sessions...) have become essential to increase patient's survival.

Withdrawal of invasive mechanical ventilation remains a daily issue and traditionally requires the transition from fully controlled ventilation to pressure support ventilation. Among specific settings of the latter, the adjustment of the trigger value (or threshold for triggering the ventilator) has not been explored to date. The trigger threshold corresponds to the sensitivity of the ventilator to detect patient's inspiratory effort and then deliver the predefined pressure support to inflate the lungs and deliver a tidal volume. The lower (or more sensitive) the trigger threshold, the smallest patient's effort will be rewarded. On the other hand, the higher the threshold, the greater the inspiratory effort required from the patient. Usually, this value is set by default to the minimum level to avoid self-triggering of the ventilator. With the objective to optimize pulmonary aeration, the use of higher trigger levels could increase diaphragmatic work (with a potential re-training and reinforcement effect) and contribute to better alveolar recruitment in the postero-inferior territories that are traditionally the most impacted, following a higher diaphragmatic motion. The authors propose to explore the impact of different trigger levels on pulmonary aeration (evaluated by electrical impedance tomography) and ventilatory parameters, in order to validate our hypotheses and before considering a trial with the objective of defining individualized trigger levels, according to patient's respiratory mechanics and pulmonary parenchyma morphology, with potential benefits on ventilator weaning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient hospitalized in the Intensive Care Unit of Clermont-Ferrand's Hospital
* Patients with mechanical invasive ventilation in spontaneous ventilation with inspiratory support (intubation or tracheostomy)
* Trigger level set to minimum
* Patient under sedation compatible with spontaneous ventilation (SV) with inspiratory support (AI) and positive end-expiratory pressure (PEP) Patient calm (RASS between -2 and 0) Consent for participation or consent from patient's next of kin or inclusion according to an emergency procedure Patient benefiting from the French social security scheme

Exclusion Criteria:

* Refusal to participate in the proposed study
* Contraindication to the installation of a nasogastric tube:

  * Severe disorder of uncorrected blood clotting
  * Known nasosinus lesion
  * Oesophageal varices recently ligated (<48h)
* Contraindication to the use of the electro-impedancemetry technique by tomography

  * Thoracic lesions
  * Chest dressings
  * Pace-maker / Implantable Defibrillator
* Known lesion of central respiratory centers, including patients with neurological injury
* Patients with Acute Respiratory Distress Syndrome (according to Berlin criteria)
* Patients with restrictive or obstructive pulmonary pathology
* Patients admitted post-operatively for surgery that may affect the diaphragmatic function ( thoracic or abdominal supra-mesocolic)
* Patients with abdominal distention (ileus, intra-abdominal hyperpressure)
* Patient whose BMI is greater than 35 kg.m-2
* Pregnant patient
* Patient under guardianship,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Lung volume (end expiratory lung volume, EELV) at each trigger level | T0 (before the first trigger step)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T15 minutes (last minute of the trigger step n°1)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T30 minutes (last minute of the trigger step n°2)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T45 minutes (last minute of the trigger step n°3)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T60 minutes (last minute of the trigger step n°4)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T75 minutes (last minute of the trigger step n°5)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T90 minutes (last minute of the trigger step n°6)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T105 minutes (last minute of the trigger step n°7)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T120 minutes (last minute of the trigger step n°8)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T135 minutes (last minute of the trigger step n°9)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol
Lung volume (end expiratory lung volume, EELV) at each trigger level | T150 minutes (last minute of the trigger step n°10)
  The main endpoint is the difference between the lung volume (EELV) measured by electroimpedancemetry by tomography (EIT) at the end of each trigger level (15th minute) and the basal value measured at the beginning of the protocol

SECONDARY OUTCOMES:
Homogeneity of pulmonary aeration | Through study completion, 150 minutes
  Evaluation of homogeneity of pulmonary aeration with Center Of Ventilation by EIT
Homogeneity of pulmonary aeration | Through study completion, 150 minutes
  Evaluation of homogeneity of pulmonary aeration with Global Inhomogeneity index by EIT
Regional impedance variation | Through study completion, 150 minutes
  Evaluation of regional impedance variation (TIV: Tidal Impedance Variation) by EIT
Atelectrauma | Through study completion, 150 minutes
  Assessement of atelectrauma (RVD: Regional Ventilation Delay) by EIT
Lung volume variations | Through study completion, 150 minutes
  Evaluation of lung volume variations by EIT (EELI : End Expiratory Lung Impedance)
Transpulmonary pressure | Through study completion, 150 minutes
  Evaluation of maximum transpulmonary pressure (alveolar stress)
Alveolar strain defined as the ratio between tidal volume and Functional Residual Capacity | Through study completion, 150 minutes
  Alveolar strain defined as the ratio between tidal volume and Functional Residual Capacity
Transpulmonary driving pressure | Through study completion, 150 minutes
  Evaluation of transpulmonary driving pressure
Work of breathing | Through study completion, 150 minutes
  Evaluation of work of breathing (WOB) value (P01)
Work of breathing | Through study completion, 150 minutes
  Evaluation of inspiratory occlusion pressure values (P01)
Energy delivered | Measurement during the last minute of each trigger step
  Evaluation of energy delivered to lungs patient
Diaphragm thickening | Through study completion, 150 minutes
  Evaluation of the diaphragmatic thickening by ultrasound
Diaphragm motion | Through study completion, 150 minutes
  Evaluation of the diaphragmatic motion by ultrasound
Patient's weight | Through study completion, 150 minutes
  Study of the impact of patient's weight

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Adultes et Soins Continus, Clermont-Ferrand, France